CLINICAL TRIAL: NCT01114386
Title: Clinical, Functional and Biological Assessment of Patients With Chronic Obstructive Pulmonary Disease (COPD) and/or Chronic Heart Failure(CHF) in Stable Conditions and During Exacerbation
Brief Title: Clinical Assessment of Patients With Chronic Obstructive Pulmonary Disease (COPD) and/or Chronic Heart Failure (CHF)
Status: Completed | Type: Observational
Sponsor: University of Modena and Reggio Emilia (Other)
Collaborators: Agenzia Italiana del Farmaco (Other Government)
Responsible Party: Principal Investigator, Leonardo M. Fabbri, Professor Medical Doctor, University of Modena and Reggio Emilia
Other Study IDs: RFPS-2006-8-334056
Record Dates: First submitted 2010-04-30; First posted 2010-05-03 (Estimated); Last update posted 2012-06-07 (Estimated); Status verified 2012-06

CONDITIONS: COPD; Heart Failure, Congestive
Keywords: Smoking; Dyspnea; Cough; Exercise
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure; Smoking; Dyspnea; Cough; Motor Activity | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sampling for routine (haemachrome and differential cells blood count, bilirubin, cholesterol, high density lipoprotein, low density lipoprotein, glycemia, blood urea, blood electrolytes (sodium, potassium, chloride), glutamic-oxaloacetic transaminase, glutamic-pyruvic transaminase, γGT, triglycerides, creatinine, uric acid, creatine phosphokinase, glycosylated haemoglobin).
  Blood sampling for selected biomarkers: NTBNP, HS-PCR and IL-6, IL1-β, cellular receptor D6 and TIR8, IL-1 decoy receptor PTX3.
  Measurement of arterial blood gases.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD patients, CHF patients: COPD and CHF patients with smoking history (> 10 pack/years), male and female, older than 50 years, referred to Hospital for dyspnea and chronic cough.
  Interventions: Procedure: Lung function testing, echocardiography, blood sampling

INTERVENTIONS:
Procedure: Lung function testing, echocardiography, blood sampling — All patients will undergo to:
  * physical examination
  * 6' Minute Walk test
  * pulmonary function testing (spirometry + volumes and reversibility testing)
  * carbon monoxide diffusing capacity (DLCO) with single-breathe technique
  * ECG
  * echocardiography

SUMMARY:
Cigarette smoking, the major risk factor for COPD, causes not only airway and lung inflammation, but also systemic effects. These systemic effects of smoking could substantially contribute to the development of chronic diseases, other than COPD, particularly chronic heart failure (CHF). The aim of this project is to assess the frequency and severity of CHF and COPD in outpatients with history of smoking referred to Hospital because of dyspnea and/or chronic cough.

DETAILED DESCRIPTION:
We will recruit 100 patients older than 50 years with diagnosis of COPD and/or CHF. COPD is defined by presence of fixed airflow obstruction (post-bronchodilator FEV1/FVC less than 70%) according to Global Initiative for Obstructive Lung Disease (GOLD) guidelines. Each patient will be characterized by medical history and physical examination. Patients with a diagnosis of COPD must have: 1) had a history of chronic respiratory symptoms, i.e., cough and sputum and/or breathlessness and only occasional wheezing (SGRQ and MMRC Questionnaire); 2) they had to be smokers or ex-smokers with more than 10 pack-years, and 3) a documented absence of a history of variable airflow obstruction and/or diagnosis of asthma. Each patient will perform pulmonary function tests, including reversibility to inhaled bronchodilator (400 µg albuterol); arterial blood gases, and routine blood tests. In addition, each patient will undergo regular PA/LL chest x-ray. The diagnosis of CHF is established according to the criteria of European Society of Cardiology. At time of entry in the study, all patients will be in clinically stable condition (ie, no changes in medication dosage or frequency, and no exacerbations of disease or hospital admissions in the preceding 6 weeks). Clinical and biological follow-up of these patients will be prospectively followed for 2 years, from 2009 to 2011.

ELIGIBILITY:
Inclusion Criteria:

* Caucasians
* Males and females
* Age > 50 years
* Smoking history > 10 pack years
* Diagnosis of COPD according to GOLD 2008 and/or diagnosis of CHF according to ESC 2008

Exclusion Criteria:

* History of bronchial asthma
* Fixed airflow limitation due to other chronic diseases such as cystic fibrosis, bronchiolitis obliterans organizing pneumonia (BOOP), bronchiectasis, TBC etc.
* Combined restrictive-obstructive functional impairment

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 patients older than 50 years with diagnosis of COPD and/or CHF, male or female, smokers or ex-smokers with more than 10 pack-years, in stable conditions.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2006-10; Primary Completion 2011-07 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo M Fabbri, MD, Principal Investigator — University of Modena and Reggio Emilia
Locations (1):
- Azienda Ospedaliero-Universitaria di Modena, Modena, Modena, Italy